CLINICAL TRIAL: NCT02086032
Title: The Effect of Different Types of Progestin on Sleeping of Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Ekachai Leeangkoonsathian, MD, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBG-2556-02070
Record Dates: First submitted 2014-03-01; First posted 2014-03-13 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Menopausal and Postmenopausal Disorders
Keywords: Sleeping quality; menopause; climacteric; progestin; dydrogesterone; micronized progesterone
MeSH Terms: interventions — Estradiol; Estrogens; Dydrogesterone; Progesterone; Utrogestan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- micronized progesterone (Experimental): 1 mg 17 beta-estradiol plus 100 mg micronized progesterone taken orally once a day for 3 months.
  Interventions: Drug: 1mg 17 beta-estradiol; Drug: micronized progesterone
- dydrogesterone (Experimental): 1mg 17 beta-estradiol plus 10 mg dydrogesterone taken orally once a day for 3 months.
  Interventions: Drug: 1mg 17 beta-estradiol; Drug: Dydrogesterone

INTERVENTIONS:
Drug: 1mg 17 beta-estradiol — Comparing sleeping quality between micronized progesterone and dydrogesterone users.
  Other Names: Estrogen
Drug: Dydrogesterone — Comparing sleeping quality between micronised progesterone and dydrogesterone users.
  Other Names: Duphaston
  Arms: dydrogesterone
Drug: micronized progesterone — Comparing sleeping quality between micronised progesterone and dydrogesterone users
  Other Names: Utrogestan
  Arms: micronized progesterone

SUMMARY:
Investigators have found that sleeping disorder is an important problem in menopausal women.

There have been papers reporting the effect of hormonal therapy on sleeping, but fews have reported the effect of different progestogens on sleeping quality. There is a need for more in-depth study and more conclusive evidence about the progestins which have the most beneficial effects on sleeping disorders in menopausal women.

This study is going to collect the data from newly identified menopausal patients who are eligible for continuous estrogen-progestogen therapy for their climacteric treatment. The affects of the therapy will be monitored for 3 months.

DETAILED DESCRIPTION:
New patients who are eligible for hormonal therapy will be selected.

They will be allocated randomly into 2 different groups, each group being prescribed 1 of 2 regimens of hormonal therapy:

* 17 beta estradiol 1mg/day plus oral micronized progesterone 100mg/day
* 17 beta estradiol 1mg/day plus dydrogesterone 10mg/day Patients will have their sleeping quality accessed using the Pittsburgh sleep quality index(PSQI) at their 1st visit and once a month for 3 months. The first and third PSQI score will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* new menopausal patients at Maharaj Nakorn Chiang Mai Hospital
* suitable for estrogen plus progesterone treatment

Exclusion Criteria:

* contraindication for hormone replacement therapy
* recently used sleep enhancing medicine
* recently used psychotic medicine

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Improving of sleeping quality (assessed by the PSQI score) | from March 2014 up to 15 months

SECONDARY OUTCOMES:
The side effects comparing the 2 arms. | from March 2014 up to 15 months
  Acne,melanoma, breast tenderness, abnormal vaginal bleeding, weight change
The climacteric symptoms comparing the 2 arms. | from March 2014 up to 15 months
  self reported of hot flash, fatigue and weakness

CONTACTS AND LOCATIONS:
Overall Officials: Tawiwan Pantasri, MD, Principal Investigator — Faculty of Medicine, Chiang Mai University, Thailand
Locations (1):
- Obstetrics and Gynecology department, Faculty of Medicine, Chiang Mai University, Muang, Chiang Mai, Thailand

REFERENCES:
- [Derived] Leeangkoonsathian E, Pantasri T, Chaovisitseree S, Morakot N. The effect of different progestogens on sleep in postmenopausal women: a randomized trial. Gynecol Endocrinol. 2017 Dec;33(12):933-936. doi: 10.1080/09513590.2017.1333094. Epub 2017 Jun 13. PMID 28609128